CLINICAL TRIAL: NCT00614094
Title: Maternal Hypoglycemia During One Hour Glucose Tolerance Test as a Risk for Decreased Placental Weight and Placental Pathology
Brief Title: Maternal Hypoglycemia and Placental Pathology
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: J. Martin Beal, Oklahoma State University Center for Health Sciences Dept. of OB/Gyn
Other Study IDs: 2007043
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Maternal Hypoglycemia
Keywords: placenta, hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this retrospective pilot study is to assess the association of maternal hypoglycemia during the one hour glucose tolerance test with decreased placental weight and identifiable placental pathology. We hypothesize that a decreased one hour glucose tolerance test is a risk factor for decreased placental weight, an increased fetal to placental weight ratio, and other identifiable placental pathology.

DETAILED DESCRIPTION:
There have been several studies linking hyperglycemia during pregnancy to adverse perinatal outcomes such as macrosomia, fetal cardiac defects, and shoulder dystocia. However, there have only been a few studies addressing the effects of hypoglycemia on perinatal outcomes. Several of these studies have shown an increased risk of intrauterine growth restriction (IUGR) with maternal hypoglycemia particularly during the glucose tolerance test (GTT).3-6 However, many of these studies have not taken into account comorbid factors or have conflicting findings.3-6 IUGR is defined as infant birth weights below the tenth percentile when the baby is otherwise genetically normal. The purpose of this retrospective pilot study is to assess the association of maternal hypoglycemia during the one hour glucose tolerance test with decreased placental weight and identifiable placental pathology. We hypothesize that a decreased one hour glucose tolerance test is a risk factor for decreased placental weight, an increased fetal to placental weight ratio, and other identifiable placental pathology.

Abell et al. found that maternal hypoglycemia during the one hour GTT was associated with decreased birth weights and intrauterine growth restriction (IUGR). However, this study made no comment on the effect of confounding factors such as tobacco use, history of gestational diabetes, or maternal BMI. Both Sokol et al and Langer et al revealed a link between decreased maternal response during the third trimester GTT and IUGR, although in the Sokol study, each pregnancy had one known risk factor for gestational diabetes. Conversely, several more recent papers have reported that maternal hypoglycemia is not predictive of IUGR or poor perinatal outcomes. -8 Consequently, the effect maternal hypoglycemia during the oral GTT is unclear. The placenta is viewed as a reflection of the intrauterine environment during pregnancy. Therefore, we wish to examine hypoglycemia during the oral one hour GTT as a risk factor for decreased placental weight, increased fetal weight to placental weight ratio, and an increased incidence of abnormal placental pathology.

A normal term placenta weighs approximately 450 grams, which is on average, one sixth of the fetal weight.9 Increased maternal substrate availability of vital fetal nutrients, such as glucose, has been known to result in large for gestational age infants, such as occurs with gestational diabetics.10 This may also be reflected in the increased placental weights linked with large for gestational age infants.11 Conversely, IUGR and small for gestational age infants may have decreased placental weights, possibly due to decreased substrate availability secondary to maternal hypoglycemia. 12 Increased fetal to placental weight ratios of 1.5 or greater above the average value for a particular gestational age are also indicative of an IUGR infant.

Identifying a possible indicator for an increased risk of decreased placental weight, which may in turn indicate an increased risk for IUGR, is vitally important when considering the outcomes of IUGR infants. These infants are at great risk for hypoglycemia, sepsis, seizure, stillbirth, respiratory distress, and meconium aspiration. Long term outcomes include poor school performance, hyperactivity, hypertension, and cardiovascular disease.2 Study Population Inclusion/Exclusion Criteria Our study population will consist of women younger than 35, who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1, 2005 and July 31, 2007. This time range was selected in order to have an adequate number of recent charts to review. (Women 35 and older are considered "advanced maternal age" and may be at increased risk of placental pathology for that reason, so they are excluded.) We expect to collect approximately 350 usable charts, with perhaps only 35 of those from patients with blood sugars in the "low" or experimental category. A power analysis using these assumptions is provided at the end of this protocol. All placentas are sent to pathology on a routine basis. A term infant is defined as delivery at 37 weeks or greater.

The study population will consist of a typical resident clinic patient population from the OSU OB-Gyn clinic. The ethnicities of the study population include African-American, Caucasian, Hispanic, American Indian, and Asian women. The population included in the study must have a one hour glucose tolerance test result equal to or less than 88 mg/dl. These results are equal to a range in the fifth percentile or less.3 We used 50 grams of oral glucola at 24 weeks or greater for our glucose tolerance test.

We will exclude women with the following comorbid conditions, due to the fact that such conditions manifest placental pathology and may affect placental weight: insufficient gestational dates, multiple gestation, hypothyroidism, hyperthyroidism, heart disease, tobacco use, drug use, history of or current gestational diabetes, history of IUGR, chromosomal abnormalities, congenital malformations, preexisting diabetes, any autoimmune disease, hypertensive disorders, abnormal maternal screen, pulmonary disease, previous gastric bypass, any disease process that results in decreased gastrointestinal absorption, HIV, intrauterine amniotic infection, history of placental abruption, thrombophilia, body mass index (BMI) greater than 40 or BMI less than 19.8.13

Early Termination Criteria N/A

Methods/Procedures Diagnosis

The diagnosis of maternal hypoglycemia after a one hour glucola screen will be defined as a one hour plasma glucose measurement of equal to or less than 88 mg/dl. The glucose screen will be performed at 24 weeks gestation or greater, as calculated by last menstrual period and ultrasound. The one hour GTT results will be obtained from the patient's chart. A decreased placental weight will be defined as a weight equal to or below one standard deviation of the mean placental weight according to gestational age (Table 1). The control group of this population will have a one hour GTT result greater than 88mg/dl. In this study, we will assess placental weight, birth weight, the placenta to birth weight ratio, and placental pathology as described in Table 2. All placental findings were assessed by a single pathologist blinded to the patient's one hour GTT results.

Data Collection The collaborating investigators and research assistants will collect age, height, weight at initial visit, date of delivery, infant birth weight, one hour GTT result, smoking and drug use status, placental weight and pathology results, and any of the above mentioned exclusion criteria only from any patient chart. (Height and weight are needed to calculate BMI.) Research assistants will be utilized to aid in the collection of this data from clinic and hospital records. These assistants will be OSU medical students employed by the work study program and will have basic human research and HIPAA training.

Analysis The two populations will be compared for various response variables. Whenever the response variable is meaningfully numeric and continuous in nature, two population t-tests will be used to compare the means of the two groups. When the response is categorical in nature, contingency tables will be created and Chi Squares tests utilized to compare the proportion of responses for the two groups. All analyses will be conducted with the use of PC SAS Version 9 (SAS Institute, Cary, NC).

Confidentiality The records reviewed will be kept in the Houston Park medical records department or Tulsa Regional Medical Center health information management department. Both these facilities are locked or under security supervision at all times. All study records will be de-identified by conversion to numbers before review, analysis, or interpretation. J. Martin Beal, D.O., Sarah McCoy, Ph.D., and Elsa Vadakekut, D.O. will have access to these numbers which will be kept locked in the OSU Ob/Gyn office, which is separate from both medical records departments. All documents linking patient names to charts will be destroyed after the data collection is complete.

ELIGIBILITY:
Inclusion Criteria:

* women younger than 35, who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1, 2005 and July 31, 2007

Exclusion Criteria:

* insufficient gestational dates, multiple gestation, hypothyroidism, hyperthyroidism, heart disease, tobacco use, drug use, history of or current gestational diabetes, history of IUGR, chromosomal abnormalities, congenital malformations, preexisting diabetes, any autoimmune disease, hypertensive disorders, abnormal maternal screen, pulmonary disease, previous gastric bypass, any disease process that results in decreased gastrointestinal absorption, HIV, intrauterine amniotic infection, history of placental abruption, thrombophilia, body mass index (BMI) greater than 40 or BMI less than 19.8

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women younger than 35, who delivered a term infant either by vaginal delivery or cesarean section at Tulsa Regional Medical Center between July 1, 2005 and July 31, 2007
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Beal, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences Dept of OB/Gyn
Locations (1):
- Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Casey BM, Lucas MJ, Mcintire DD, Leveno KJ. Pregnancy outcomes in women with gestational diabetes compared with the general obstetric population. Obstet Gynecol. 1997 Dec;90(6):869-73. doi: 10.1016/s0029-7844(97)00542-5. PMID 9397092
- [Background] Abell DA, Beischer NA. Evaluation of the three-hour oral glucose tolerance test in detection of significant hyperglycemia and hypoglycemia in pregnancy. Diabetes. 1975 Oct;24(10):874-80. doi: 10.2337/diab.24.10.874. PMID 1175859
- [Background] Sokol RJ, Kazzi GM, Kalhan SC, Pillay SK. Identifying the pregnancy at risk for intrauterine growth retardation: possible usefulness of the intravenous glucose tolerance test. Am J Obstet Gynecol. 1982 May 15;143(2):220-3. doi: 10.1016/0002-9378(82)90658-5. PMID 7081335
- [Background] Langer O, Damus K, Maiman M, Divon M, Levy J, Bauman W. A link between relative hypoglycemia-hypoinsulinemia during oral glucose tolerance tests and intrauterine growth retardation. Am J Obstet Gynecol. 1986 Oct;155(4):711-6. doi: 10.1016/s0002-9378(86)80004-7. PMID 3532796
- [Background] Calfee EF, Rust OA, Bofill JA, Ross EL, Morrison JC. Maternal hypoglycemia: is it associated with adverse perinatal outcome? J Perinatol. 1999 Jul-Aug;19(5):379-82. doi: 10.1038/sj.jp.7200048. PMID 10685261
- [Background] Weissman A, Solt I, Zloczower M, Jakobi P. Hypoglycemia during the 100-g oral glucose tolerance test: incidence and perinatal significance. Obstet Gynecol. 2005 Jun;105(6):1424-8. doi: 10.1097/01.AOG.0000159577.28448.f9. PMID 15932839
- [Background] Feinberg JH, Magann EF, Morrison JC, Holman JR, Polizzotto MJ. Does maternal hypoglycemia during screening glucose assessment identify a pregnancy at-risk for adverse perinatal outcome? J Perinatol. 2005 Aug;25(8):509-13. doi: 10.1038/sj.jp.7211336. PMID 15908987